CLINICAL TRIAL: NCT05656196
Title: To Evaluate the Chinese Herbal Tea VGH-DESJS-1 in Ocular and Oral Dryness Symptoms of Dry Eye Syndrome and Sjögren's Syndrome
Brief Title: VGH-DESJS-1 in Ocular and Oral Dryness Symptoms of Dry Eye Syndrome and Sjögren's Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022-08-011A
Record Dates: First submitted 2022-08-09; First posted 2022-12-19 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Dry Eye Syndrome; Sjogren's Syndrome; Xerophthalmia
Keywords: Dry Eye Syndrome; Sjogren's Syndrome; Xerophthalmia; Chinese herbal tea; Nourishing Yin and Moistening Dryness
MeSH Terms: conditions — Dry Eye Syndromes; Sjogren's Syndrome; Xerophthalmia

STUDY DESIGN:
Intervention Model Description: 30 dry eye syndrome subjects, 60 Sjögren's syndrome' dry eye subjects, and 10 non DES SJS Healthy Controls, NHC)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dry eye syndrome (DES) (Experimental): Dry eye syndrome (DES) will received Chinese herbal tea VGHTPE-DESJS-1 8 weeks on Nourishing Yin and Moistening Dryness the ocular dryness evaluation. And we could use the Schirmer's test, Tear breakup time, Ocular Surface Disease Index (OSDI), EULAR Sjogren's Syndrome Patient Reported Index (ESSPRI), Pittsburgh Sleep Quality Index (PSQI), Ford Insomnia Response to Stress Test (FIRST), cytokine markers, Whole-genome genotyping, TCM pattern, Traditional Chinese Medicine (TCM) tongue diagnosis, TCM pulse diagnosis, and TCM heart rate variability for this purpose.
  Interventions: Other: Chinese herbal tea VGH-DESJS-1
- Sjögren's syndrome (SJS) (Experimental): Sjögren's syndrome (SJS) will received Chinese herbal tea VGHTPE-DESJS-1 8 weeks on Nourishing Yin and Moistening Dryness the ocular dryness evaluation. And we could use the Schirmer's test, Tear breakup time, Ocular Surface Disease Index (OSDI), EULAR Sjogren's Syndrome Patient Reported Index (ESSPRI), Pittsburgh Sleep Quality Index (PSQI), Ford Insomnia Response to Stress Test (FIRST), cytokine markers, Whole-genome genotyping, TCM pattern, Traditional Chinese Medicine (TCM) tongue diagnosis, TCM pulse diagnosis, and TCM heart rate variability for this purpose.
  Interventions: Other: Chinese herbal tea VGH-DESJS-1
- Non DES SJS Healthy Controls (NHC) (Experimental): Non DES SJS Healthy Controls (NHC) will received Chinese herbal tea VGHTPE-DESJS-1 8 weeks on Nourishing Yin and Moistening Dryness the ocular dryness evaluation. And we could use the Schirmer's test, Tear breakup time, Ocular Surface Disease Index (OSDI), EULAR Sjogren's Syndrome Patient Reported Index (ESSPRI), Pittsburgh Sleep Quality Index (PSQI), Ford Insomnia Response to Stress Test (FIRST), cytokine markers, Whole-genome genotyping, TCM pattern, Traditional Chinese Medicine (TCM) tongue diagnosis, TCM pulse diagnosis, and TCM heart rate variability for this purpose.
  Interventions: Other: Chinese herbal tea VGH-DESJS-1

INTERVENTIONS:
Other: Chinese herbal tea VGH-DESJS-1 — Chinese herbal tea VGH-DESJS-1.

SUMMARY:
To evaluate the Chinese herbal tea VGH-DESJS-1 in ocular and oral dryness symptoms of Dry eye syndrome and Sjögren's syndrome

DETAILED DESCRIPTION:
Method: This study wants to evaluate the Chinese herbal tea VGH-DESJS-1 on Nourishing Yin and Moistening Dryness the ocular dryness from dry eye syndrome (DES) and Sjögren's syndrome (SJS). One hundred dry eye subjects are composed of 30 dry eye syndrome subjects, 60 Sjögren's syndrome' dry eye subjects, and 10 non DES SJS Healthy Controls, NHC). DES, SJS, and NHC received VGH-DESJS-1 daily during 8 weeks for the evaluation before and after the subjects receiving the VGH-DESJS-1. Moreover, we could use the Whole-genome genotyping, Schirmer's test, Tear breakup time (TBUT), Cytokines, Ocular Surface Disease Index (OSDI), EULAR Sjogren's Syndrome Patient Reported Index (ESSPRI), Pittsburgh Sleep Quality Index (PSQI), Ford Insomnia Response to Stress Test (FIRST), Traditional Chinese Medicine (TCM) pattern, TCM tongue diagnosis, TCM pulse diagnosis, and TCM heart rate variability, and it could be applied for the goal of holistic health care.

Expected Results:

1. To evaluate the difference among Schirmer's test, TBUT, TCM pattern, TCM tongue diagnosis, TCM pulse diagnosis, heart rate variability, Whole-genome genotyping, and Cytokines for DES, SJS, and NHC.
2. To evaluate the Nourishing Yin and Moistening Dryness of VGH-DESJS-1 for DES and SJS.
3. To evaluate the Nourishing Yin and Moistening Dryness of VGH-DESJS-1 for DES.
4. To evaluate the Nourishing Yin and Moistening Dryness of VGH-DESJS-1 for SJS.

Keywords: Dry eye syndrome, Sjögren's syndrome, Xerophthalmia, Chinese herbal tea, Nourishing Yin and Moistening Dryness

ELIGIBILITY:
Dry eye syndrome

-Inclusion Criteria: aged between 20 and 75 years Schirmer's test less than 10 mm/5 min

-Exclusion Criteria: Pregnancy With eye inflammation or infectious eye disease Accepted operation of eye

Sjögren's syndrome

-Inclusion Criteria: primary or secondary SS aged between 20 and 75 years fulfilled the 2002 American-European Consensus Criteria for SS (AECG) had no abnormal findings of immune, liver, kidney, or blood function evaluations.

-Exclusion Criteria: a history of alcohol abuse, diabetes mellitus, or major life-threatening condition pregnancy or breastfeeding steroid pulse therapy within three months prior to the commencement of our study.

non AIDDES Healthy Controls

-Inclusion Criteria: aged between 20 and 75 years without any Chronic disease

-Exclusion Criteria: any Sjögren's syndrome or Dry eye syndrome.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Schirmer's test | 8 weeks
  Dry eye syndrome (DES) and Sjögren's syndrome (SJS) take the Schirmer's test.
Ocular Surface Disease Index (OSDI) | 8 weeks
  Dry eye syndrome (DES) and Sjögren's syndrome (SJS) take the OSDI(Ocular Surface Disease Index).

SECONDARY OUTCOMES:
TCM pattern | 8 weeks
  Dry eye syndrome (DES), Sjögren's syndrome (SJS), and on DES SJS Healthy Controls (NHC) take the TCM pattern to differentiate the 9 types of TCM constitutions.
TCM tongue diagnosis | 8 weeks
  Dry eye syndrome (DES), Sjögren's syndrome (SJS), and on DES SJS Healthy Controls (NHC) take the TCM tongue diagnosis with camera photo to differentiate the TCM tongue feature factors about Tongue body, Tongue Coating, Red spot, Tooth marks, and Ecchymosis. TCM tongue feature factors would present the status of inflammation, blood stasis, heat, dampness with TCM theory.
TCM pulse diagnosis | 8 weeks
  Dry eye syndrome (DES), Sjögren's syndrome (SJS), and on DES SJS Healthy Controls (NHC) take the TCM pulse diagnosis with blood pressure monitors to differentiate the TCM pulse feature factors about Floating, Deep, Slow, Rapid, Deficient, Excessive, Slippery, Rough, String-like, Soggy, Fine, Weak. TCM tongue feature factors would present the status of inflammation, blood stasis, heat, dampness with TCM theory.
TCM heart rate variability | 8 weeks
  Dry eye syndrome (DES), Sjögren's syndrome (SJS), and on DES SJS Healthy Controls (NHC) take the TCM heart rate variability.
Whole-genome genotyping(TWBv2.0) | 8 weeks
  Dry eye syndrome (DES), Sjögren's syndrome (SJS), and on DES SJS Healthy Controls (NHC) take the Whole-genome genotyping (TWBv2.0).
Cytokine markers | 8 weeks
  Dry eye syndrome (DES), Sjögren's syndrome (SJS), and on DES SJS Healthy Controls, NHC) take the cytokine markers (IL-17, MMP-9, BAFF, BCMA) analysis.
Pittsburgh Sleep Quality Index | 8 weeks
  Dry eye syndrome (DES), Sjögren's syndrome (SJS), and on DES SJS Healthy Controls, NHC) take the Pittsburgh Sleep Quality Index
Ford Insomnia Response to Stress Test | 8 weeks
  Dry eye syndrome (DES), Sjögren's syndrome (SJS), and on DES SJS Healthy Controls, NHC) take the Ford Insomnia Response to Stress Test.
EULAR Sjogren's Syndrome Patient Reported Index (ESSPRI) | 8 weeks
  Dry eye syndrome (DES), Sjögren's syndrome (SJS), and on DES SJS Healthy Controls, NHC) take the EULAR Sjogren's Syndrome Patient Reported Index (ESSPRI)

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Mao Chang, M.D., Ph.D., Principal Investigator — Center for Traditional Medicine, Taipei Veterans General Hospital, Taipei, Taiwan
Locations (1):
- Ching-Mao Chang, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No